CLINICAL TRIAL: NCT00024310
Title: A Phase I Trial of Lometrexol Sodium and Paclitaxel Adminsitered Intravenously Every 21 Days in Conjunction With Oral Folic Acid in Patients With Solid Tumors
Brief Title: Paclitaxel, Folic Acid, and Lometrexol in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068917; UCLA-0005068; TULA-T3004; NCI-G01-2017
Record Dates: First submitted 2001-09-13; First posted 2003-06-20 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2002-11

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; drug/agent toxicity by tissue/organ
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Folic Acid; lometrexol; Paclitaxel

INTERVENTIONS:
Dietary Supplement: folic acid
Drug: lometrexol
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Folic acid may protect normal cells from the side effects of chemotherapy and may increase the effectiveness of chemotherapy by making tumor cells more sensitive to the drug. Lometrexol may stop the growth of tumors by blocking one of the enzymes necessary for cancer cell growth. Combining chemotherapy with folic acid and lometrexol may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining paclitaxel, folic acid, and lometrexol in treating patients who have locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II study dose of lometrexol and paclitaxel when combined with folic acid in patients with locally advanced or metastatic solid tumors.
* Determine the quantitative and qualitative toxic effects of this regimen in these patients.
* Determine the plasma concentrations of lometrexol and paclitaxel and relate their pharmacokinetics to toxicity outcome in these patients.
* Determine the antitumor activity of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of lometrexol and paclitaxel.

Patients receive lometrexol IV over 30-60 seconds immediately followed by paclitaxel IV over 3 hours on day 1. Patients also receive oral folic acid beginning 7 days before lometrexol/paclitaxel and continuing for 14 days. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Doses of lometrexol and paclitaxel are escalated sequentially. Cohorts of 3-6 patients receive escalating doses of lometrexol and paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 6 patients experience dose-limiting toxicity. Six to twelve additional patients are treated at the recommended phase II study dose (dose immediately preceding the MTD).

Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 12-42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven locally advanced or metastatic solid tumor that is refractory to standard therapies or for which there are no therapies of potential major benefit
* Measurable disease
* No hematologic malignancies, including leukemia, lymphoma, or multiple myeloma
* No symptomatic effusions or ascites unless drained before study entry
* No clinically apparent CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3*
* Platelet count at least 100,000/mm^3*
* Hemoglobin at least 9.0 g/dL* NOTE: * Without growth factor support

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT and SGPT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if tumor involvement of liver)
* Albumin greater than 2.5 g/dL

Renal:

* Glomerular filtration rate at least 65 mL/min

Gastrointestinal:

* No inflammatory bowel disease
* No radiation enteritis
* No malabsorption syndrome

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to study drugs or related compounds (e.g., LY309887, multi-targeted antifolate, AG-2034, methotrexate, docetaxel, or polyoxyethylated castor oil)
* No active uncontrolled infection unless approved by the investigator
* No other severe concurrent disease that would preclude study therapy
* No body surface area greater than 3.0 m^2
* No known vitamin B12 deficiency

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent routine or prophylactic filgrastim (G-CSF), sargramostim (GM-CSF), or epoetin alfa
* No concurrent biologic-response modifiers

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin, carboplatin, or nitrosourea) and recovered
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* Recovered from prior radiotherapy
* No prior radiotherapy to 25% or more of bone marrow (e.g., whole-pelvic irradiation)
* No concurrent radiotherapy (including palliative radiotherapy)

Surgery:

* At least 4 weeks since prior major surgery and recovered

Other:

* At least 4 weeks since prior investigational agent
* No more than 2 prior therapies for locally advanced or metastatic solid tumor
* No other concurrent investigational agent
* No concurrent trimethoprim, co-trimoxazole, proguanil, or pyrimethamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Rosen, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States